CLINICAL TRIAL: NCT01927471
Title: Nutritional and Metabolic Correlates of Ovarian Morphology in Women With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: IRB #: 1108002383
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Menstrual Irregularity
Keywords: Menstrual cycles; Ultrasound; Ovary; Polycystic Ovary Syndrome (PCOS); Physical activity; Diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood serum, subcutaneous fat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Regular menstrual cycles: Adult women will be assigned to this category if they report a history of regular menstrual cycles. We will aim to recruit 120 women in this category.
- Irregular menstrual cycles, no PCOS: Adult women will be assigned to this category if they report a history of irregular menstrual cycles, without a pre-existing diagnosis of PCOS. We will aim to recruit 120 women in this category.
- Irregular menstrual cycles, with PCOS: Adult women will be assigned to this category if they report a history of irregular menstrual cycles with a pre-existing diagnosis of PCOS by a physician. We will aim to recruit 120 women in this category.

SUMMARY:
The investigators would like to determine how aspects of metabolism and age influence ovarian function. The purpose of the study is to understand how nutrition and metabolism relate to follicle development in women with regular cycles, irregular cycles, or polycystic ovary syndrome (PCOS). We also plan to identify lifestyle factors associated with PCOS and understand how diet and activity levels impact features of PCOS.

DETAILED DESCRIPTION:
In the ovaries, eggs rest in fluid filled sacs called follicles. When follicles grow they form small fluid-filled cysts that can be easily seen when we use ultrasound to view the ovaries. In women with regular menstrual cycles, groups of follicles grow and regress 2 to 3 times during their cycle (usually over a 28- day period). Several of these follicles grow to a stage where they begin to develop the potential to ovulate - but in general only one follicle is chosen to ovulate. Thus, at any given time during the menstrual cycle, numerous fluid-filled follicles can be visualized in a woman's ovaries at various stages of development using transvaginal ultrasonography. In women with absent or infrequent menstrual cycles, very little is known about the growth patterns of their follicles and how factors such as metabolic hormones, might play a role in the failure to ovulate. Being underweight or overweight increases your chances of having irregular or absent menstrual cycles and a history of abnormal reproductive function compounds your risks for chronic diseases such as infertility, diabetes, hypertension, atherosclerosis and certain cancers. This is particularly the case for women with PCOS that have menstrual cycles that appear to worsen or improve depending on their body weight and metabolic status. Polycystic ovary syndrome (PCOS) is an endocrine disorder that affects 6-12% of reproductive-aged women within the general population. The hallmark features of PCOS are menstrual irregularity, increased levels of androgens, and polycystic ovaries. The current diagnostic criteria require 2 out of 3 of these features to be present for the diagnosis, therefore a number of phenotypes of PCOS exist. However, the metabolic and reproductive differences across the phenotypic spectrum of PCOS are not well understood. Women with PCOS characteristically have polycystic ovaries, where up to 10 times more follicles are present in the ovary at any given time. Further, the follicle-size populations and overall distribution throughout the ovary varies in women - follicles may be situated around the periphery of the ovary or may be distributed throughout the ovary. Presumably these small follicles are arrested in development - but emerging data from the Lujan laboratory suggest that this is not the case. Rather, follicles continue to grow in a dynamic pattern during these prolonged periods of anovulation. By comparing follicle populations, reproductive hormones and markers of metabolism in women with regular cycles, women with irregular cycles, and women with a history of PCOS, the researchers plan to identify what factors might explain why fertility potential and long-term health are compromised in some women but not in others. By including women at both early and late stages of their reproductive potential, the researchers will also be able to assess what influence age has on these factors. The ultimate goal of this research is to understand how nutrition and metabolism regulate follicle development in women so we can better develop lifestyle and drug therapies to help women preserve their fertility and long-term health. Since obesity has recently become the leading cause of infertility in North America, these studies are especially important.

Current research has failed to thoroughly examine the relationships between dietary intake, energy expenditure and PCOS. The purpose of this proposed study is to identify lifestyle factors associated with PCOS. Through dietary intake and energy expenditure data, the researchers plan to examine potential lifestyle differences between PCOS and healthy women, as well as between BMI classifications within women with PCOS. The Research Team will also be able to evaluate the diet quality according to the USDA Dietary Guidelines for Americans of all women included in the study. The Research Team is also interested in the relationships between biological markers and lifestyle endpoints in women with and without PCOS. Previous literature has shown there are biological marker differences between those with and without PCOS. By examining these relationships, researchers may further understand whether PCOS status is associated with lifestyle parameters.

To accomplish these objectives, the investigators plan to recruit 120 women with regular menstrual cycles and 240 women with irregular menstrual cycles, with or without PCOS (sub-grouped into 120 women with irregular menstrual cycles and 120 women with a history of PCOS). Their goal is to recruit an equal number of women in each group such that they are matched for age (18 - 48 years old) and body mass index (BMI; Normal weight = 18 - 24.9 kg/m2; Overweight = 25 - 29.9 kg/m2; Obese ≥ 30kg/m2). Women will be included in the PCOS sub-group if they have a confirmed PCOS diagnosis from their primary care provider. Ultrasound scans of the ovaries will be assessed for the total number, size, and distribution of follicles using both two- and three-dimensional imaging techniques. Participants will have blood samples collected determine serum concentrations of luteinizing hormone (LH), follicle stimulating hormone (FSH), estradiol, progesterone, anti-müllerian hormone (AMH), and inhibin B. The following metabolic parameters will be assessed: (1) 75-gram oral glucose tolerance test to characterize glucose and insulin dynamics at 0, 30, 60, 90, and 120 minutes post-glucose ingestion; (2) dual X-ray absorptiometry (DXA) scan to quantify body fat and lean muscle distribution; (3) vitals and anthropometry assessment to measure waist and hip circumference, height, weight, blood pressure, and heart rate, and (4) fasting blood tests to detect serum concentrations of androgens (i.e., total testosterone, androstenedione, free androgen index) and serum markers of metabolic syndrome (i.e., lipids and hemoglobin A1C). Participants will complete a food frequency questionnaire, a semi-structured dietary interview, and physical activity questionnaire. A researcher may also provide participants with an accelerometer to wear for a week. Participants may also elect to participate in an optional subcutaneous fat biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 48 years
* BMI ≥ 18 kg/m2

Either:

* Regular menstrual cycles (21-35 days);
* Irregular menstrual cycles (>36 days); or
* Previous diagnosis of PCOS from a primary care provider
* If 21 years of age or older, must have had a healthy pelvic exam w/in the past 2 years

Exclusion Criteria:

* Current use of medication(s) known or suspected to interfere with reproductive function (eg. oral contraceptives) or insulin sensitivity
* Pregnant or breastfeeding
* Not otherwise healthy
* Significant weight changes within the last three months

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women must be able to transport to Cornell University and University of Rochester. Eligible participants are between 18-48 years with a BMI of 18 kg/m2 or higher. Women are screened and enrolled following consent based on their response to our advertisements. Enrollment is restricted to the geographical area.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2011-09; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Follicle number per ovary | 1 day
  The number and size of all follicles in each ovary will be assess by ultrasonography for each participant with regular menstrual cycles, irregular menstrual cycles and PCOS.
Insulin sensitivity | 1 day
  Insulin sensitivity will be determined by administration of an oral glucose tolerance test and compared across groups.

SECONDARY OUTCOMES:
Ovarian Volume | 1 day
  The size of each ovary will be determined by ultrasonography for each participant and compared across groups.
Anti-Müllerian hormone | 1 day
  Circulating AMH levels in the serum will be determined for each participant and compared across groups.
LH-FSH ratio | 1 day
  The ratio of circulating LH to FSH concentrations in the serum will be determined for each participant and compared across groups.
Androgen concentrations | 1 day
  Total testosterone, androstenedione and free androgen index concentrations in serum will be determined and compared across groups.
Menstrual Cycle Length | 1 day
  Average menstrual cycle length as determined by self-reported history will be determined and compared across groups.
Hirsutism | 1 day
  Degree of hirsutism as judged by the Ferriman-Gallwey scale will be determined and compared across groups.
Serum markers of metabolic syndrome | 1 day
  Lipids, glucose and HbA1C concentrations will be determined and compared across groups.
Blood Pressure | 1 day
  Blood pressure will be determined and compared across groups.
Body mass index | 1 day
  The ratio of weight to height will be determined and compared across groups.
Waist-to-hip ratio | 1 day
  The ratio of waist circumference to hip circumference will be determined and compared across groups.
Body fat distribution | 1 day
  Percentage and distribution of fat and lean mass as assessed using DXA technology will be compared across groups.
Differences in diet composition between women with and without PCOS | 1 week
  A food frequency questionnaire will be administered to assess diet composition for the last three months
Differences in energy expenditure between women with and without PCOS | 1 week
  Participants will be asked to wear a small accelerometer device to assess physical activity
Subcutaneous fat biopsy (optional) | 1 day
  Subcutaneous fat biopsies will be conducted to assess differences in fat cell populations (major site of reproductive hormone synthesis) between groups

CONTACTS AND LOCATIONS:
Overall Officials: Marla E. Lujan, PhD, Principal Investigator — Cornell University
Locations (3):
- United States (3):
  - Human Metabolic Research Unit, Cornell University, Ithaca, New York
  - Strong Fertility Center, Rochester, New York
  - CRC at University of Rochester Medical Center, Rochester, New York